CLINICAL TRIAL: NCT00815282
Title: Immune Response After Human Papillomavirus Vaccination in Patients With Autoimmune Disease
Acronym: HPV-kind
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: N.M. Wulffraat (Other)
Collaborators: National Institute for Public Health and the Environment (RIVM) (Other Government)
Responsible Party: Sponsor-Investigator, N.M. Wulffraat, MD, UMC Utrecht
Organization: UMC Utrecht (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL26.113.000.08; EUDRACT number 2008-008169-36
Record Dates: First submitted 2008-12-24; First posted 2008-12-29 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Juvenile Idiopathic Arthritis; Systemic Lupus Erythematosus; Juvenile Dermatomyositis
MeSH Terms: conditions — Arthritis, Juvenile; Lupus Erythematosus, Systemic; Dermatomyositis | interventions — Papillomavirus Vaccines; human papillomavirus vaccine, L1 type 16, 18; halofantrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients (Other): patients were girls aged 15 to 18 immunised with the HPV vaccine according to dutch vaccination guidelines
  Interventions: Other: Human papilloma virus vaccine (cervarix)

INTERVENTIONS:
Other: Human papilloma virus vaccine (cervarix) — vaccination at 0, 1 and 6 months
  Other Names: Cervarix vaccine (GlaxoSmithKLine)

SUMMARY:
In the Netherlands, the human Papillomavirus (HPV) vaccination will be added to the National Vaccination Program for girls to protect against the development of cervical cancer. The vaccine protects against HPV type 16 & 18, which cause about 75% of cervical cancer. Studies have shown that the vaccine is effective in healthy subjects in preventing infection by HPV 16 & 18. However, no evidence exists on the immunogenicity and safety of HPV vaccination in patients with an immune system disorder, such as primary humoral immunodeficiency (i.e. hypogammaglobulinemia) or autoimmune diseases. Concerns exist that vaccination may cause an aggravation of the underlying disease. In addition, the immune response to vaccination may be diminished due to immunosuppressive therapy or the underlying disease.

Objective: The primary goal of the current study is to study the immunogenicity of HPV vaccination in patients with an autoimmune disease and a primary humoral immunodeficiency.

Based on retrospective analysis with other vaccines we hypothesize that patients with autoimmune diseases who are under immunosuppressive medication and patients with a immune system disorder have a decreased serological response to HPV vaccination, and that the produced HPV antibodies titers decrease more rapidly than in healthy individuals.

The secondary objective is to explore safety of HPV vaccination and immune regulatory mechanisms induced by vaccination in a subset of patients. The investigators hypothesize that HPV vaccination is safe and that HPV-induced regulatory T cells are able to prevent an increase in the activity of an autoimmune disease.

DETAILED DESCRIPTION:
Study design: prospective observational cohort study.

Study population: Females aged 12 - 18 years with one of the autoimmune diseases Juvenile Idiopathic Arthritis (JIA), Systemic Lupus Erythematosus (SLE) and Juvenile Dermatomyositis (JDM) are included. Included females are treated at the rheumatology unit from the University Medical Center Utrecht. A small control group of healthy girls aged 13 -17 years will also be included to compare the kinetics of HPV serology with healthy individuals.

Intervention: Starting from September 2009 all girls aged 12 years will be offered a HPV vaccination via the National Vaccination Program. Prior to this, a national campaign will be started in March 2009 to vaccinate all girls aged 13-17 years at once.We will use this national vaccination campaign as an opportunity to analyze the serological response and safety of this vaccine in a large group of with an immune system disorder. The vaccines are administered by our national health organisation. The effects are monitored in our clinics.

Main study parameters/endpoints:

* Primary outcome immunogenicity is measured by antibody levels against HPV serotype 16 & 18 over time. We consider HPV vaccination to be immunogenic at antibody titers above the cutoffs 20 and 24 mMU/ml for HPV 16 and 18, respectively; or at a ≥2 fold increase in antibody levels against both serotypes. The antibody levels will be measured prior to vaccination, and after 3,7 and 12 months.
* The secondary outcome is safety of vaccination, measured as activity of the underlying autoimmune disease. In addition, frequency of common adverse effects, and immunological changes induced by HPV vaccination, such as number and function of cytotoxic T cells and Tregs will be described.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

Burden: included patients will be asked to visit the hospital 4 times in a period of 12 months. During these visits, physical examination will be performed and blood will be obtained for serological and immunological analysis. Most of these visits are combined with routine follow-up and venous punctures of the patients. However, one extra visit to the hospital and vena puncture is expected. 5 ml (extra) blood is obtained four times from all patients for serological analysis. Included healthy controls will be asked to visit one plenary information meeting in the evening. Controls will have a venous punctures four times during the study, during which 5 ml of blood is obtained. These samples will be obtained at the hospital during evening clinics or at school. In a subset of patients (n=50) and healthy controls (n=10), an additional 15 ml is obtained for immunological analysis.

Risks: participants may experience adverse events of the HPV vaccination. Benefits: Protection against human Papillomavirus infection and therefore reduced risk of cervix carcinoma, certainty about protection against HPV 16 & 18 and about safety of HPV vaccination.

Group relatedness: This study can only be done in patients who need this vaccination (i.e. females in the age group 12-24 years) and have an immune system disorder, such as JIA, SLE or JDM. Appropriate comparison with healthy controls must be performed in age-matched healthy females who are also recruited for the National HPV vaccination campaign, in this case girls in the age group 13-17 years.

ELIGIBILITY:
Inclusion Criteria:

* Females
* Clinical diagnosis of JIA, SLE or JDM
* And who are in the following age groups:

  * 12 years (these girls are vaccinated via the National Vaccination Program from September 2009)
  * 13-18 years (these girls are vaccinated during a national vaccination campaign from March-May 2009)
* Current co-medication: all co-medication prescribed may be continued
* And in the control group: healthy girls aged 13-17 years (these girls are vaccinated during a national vaccination campaign from March-May 2009)

Exclusion Criteria:

* No HPV vaccination
* Refusal to allow venous puncture
* Proven or suspected cervical carcinoma

Ages: 12 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 135 (Actual)
Dates: Start 2009-02; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
the immunogenicity of HPV vaccination in patients with immune system disorders. The immunogenicity of HPV vaccination in patients will be compared to healthy controls, measured by antibody levels against HPV serotype 16 & 18. | 0, 3, 7, 12 months

SECONDARY OUTCOMES:
difference in the activity of underlying disease before versus after vaccination. A difference in the activity of underlying autoimmune disease, will be measured according to specific criteria for each autoimmune disease. | 0,3,7,12 months

CONTACTS AND LOCATIONS:
Overall Officials: Nico M Wulffraat, MD, PhD, Principal Investigator — UMC Utrecht; Fiona van der KLis, MD, PhD, Study Director — National Institute for Public Health and the Environment; Guy Berbers, PhD, Study Director — National Institute for Public Health and the Environment
Locations (3):
- Netherlands (3):
  - University Medical center Groningen, Groningen
  - Erasmus Medical Center Rotterdam, Rotterdam
  - UMC Utrecht, department of pediatrics, Utrecht

REFERENCES:
- [Result] Heijstek MW, Pileggi GC, Zonneveld-Huijssoon E, Armbrust W, Hoppenreijs EP, Uiterwaal CS, Kuis W, Wulffraat NM. Safety of measles, mumps and rubella vaccination in juvenile idiopathic arthritis. Ann Rheum Dis. 2007 Oct;66(10):1384-7. doi: 10.1136/ard.2006.063586. Epub 2007 Feb 6. PMID 17284544
- [Result] Zonneveld-Huijssoon E, Ronaghy A, Van Rossum MA, Rijkers GT, van der Klis FR, Sanders EA, Vermeer-De Bondt PE, Hoes AW, van der Net JJ, Engels C, Kuis W, Prakken BJ, Van Tol MJ, Wulffraat NM. Safety and efficacy of meningococcal c vaccination in juvenile idiopathic arthritis. Arthritis Rheum. 2007 Feb;56(2):639-46. doi: 10.1002/art.22399. PMID 17265499
- [Result] Heijstek MW, Scherpenisse M, Groot N, Tacke C, Schepp RM, Buisman AM, Berbers GA, van der Klis FR, Wulffraat NM. Immunogenicity and safety of the bivalent HPV vaccine in female patients with juvenile idiopathic arthritis: a prospective controlled observational cohort study. Ann Rheum Dis. 2014 Aug;73(8):1500-7. doi: 10.1136/annrheumdis-2013-203429. Epub 2013 May 30. PMID 23723319